CLINICAL TRIAL: NCT03633071
Title: Prospective Trial of the TriFit™ Web Knee Brace: An Evaluation of Functional Improvements and Satisfaction in Conservatively-Managed Patients With Knee Osteoarthritis Over a 12-month Period
Brief Title: Prospective Trial of the TriFit™ Web Knee Brace
Status: Terminated | Type: Observational
Why Stopped: Low enrollment
Sponsor: Foundation for Orthopaedic Research and Education (Other)
Collaborators: DJO Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: JS - Trifit -001
Record Dates: First submitted 2017-11-07; First posted 2018-08-16 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Web-knee brace — Web -Knee Brace

SUMMARY:
This is a prospective trial comparing improvements in pain, function, and quality of life in patients with early-stage knee osteoarthritis conservatively managed with the TriFit™ Web Knee Brace. The study design will represent a consecutive series of conservatively managed patients with knee-pain not yet candidates for surgical intervention and is non-comparative in nature.

DETAILED DESCRIPTION:
This clinical study will be conducted at the Florida Orthopaedic Institute (FOI) beginning in 2017. The trial will be a prospective trial of a convenience sample of skeletally mature patients with knee pain treated by the Principal Investigator (Jeff Sellman, MD) at Florida Orthopaedic Institute with clinically and radiographically confirmed early stage knee Osteoarthritis that can be managed without surgical intervention. The study population will be defined as all adult patients (>21 years) seen by the Principal Investigator and diagnosed with knee osteoarthritis. All patients will be independent in activities of daily living. All patients will be seen in the Prinicpal Investigator outpatient clinic at Florida Orthopaedic Institute. Patients will be screened as candidates for enrollment into the study and if the patient satisfies the inclusion/exclusion criteria, a clinical research coordinator or the study Principal Investigator will explain all essential elements of the clinical trial. If the patient agrees to participate, the study coordinator or Principal Investigator will obtain informed consent. The patient will still be followed clinically for 12 months after initial brace application.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 21 years;
2. BMI < 40;
3. Medial or lateral knee Osteoarthritis as clinical diagnosis [Kellgren-Lawrence grades 1-3 Osteoarthritis];
4. Persistent knee pain beyond current treatment;
5. No history of corticosteroid injection or viscosupplementation injections in the last 3 months;
6. Able to comply with study requirements;
7. Capable and willing of signing informed consent.

Exclusion Criteria:

1. Age < 21 years;
2. History of diabetic neuropathy;
3. History of traumatic onset of knee pain;
4. Undergone surgery on either lower limb within 6 months;
5. Unable to comply with study requirements;
6. Had previously received corticosteroid injections or viscosupplementation injections in the affected knee within 3 months of study;
7. KL grade >3

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be defined as all adult patients (>21 years) seen by the Principal Investigator and diagnosed with knee osteoarthritis. All patients will be seen in the Principal Investigator's outpatient clinic at Florida Orthopaedic Institute. The patient will still be followed clinically for 12 months after initial brace application and per the schedule of assessments as described below.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score | up to12 months
  - The KOOS Jr. survey is a self-reported questionnaire (7 questions) designed to measure "knee health" as it reflects aspects of pain, symptom severity, and activities of daily living (ADL) including movement or activities that are directly relevant and difficult for patients with knee OA. A short-form knee arthroplasty outcomes survey.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) (measures pain) | Baseline (screening) and compare at specific timepoints until 12 months
  - A short-form to measure pain level knee arthroplasty outcomes survey. The scale is from 1-100 on a 10cm ruler, the higher the number equals more pain.
Activity Restriction Scores | up to12 month period
  -A scale from 1-100, 1 being no activity, and 100 being active
Patient Satisfaction with Brace | up to 12 month course of study
  Satisfaction is measured by 5 choices, very dissatisfied, dissatisfied, not dissatisfied or satisfied, satisfied, very satisfied.
Analgesic use | up to12 month course of the study
  Analgesic use for Knee pain, medications, Injections - to document subjects pain
Compliance | up to 12 month course of the study
  Compliance - to document how many hours the brace is worn

CONTACTS AND LOCATIONS:
Overall Officials: Jeff E Sellman, MD, Principal Investigator — Florida Orthopaedic Institute
Locations (1):
- Florida Orthopaedic Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
Outcomes of IPD